CLINICAL TRIAL: NCT06265701
Title: Decreasing Depressive Symptoms Through a Derailment-Focused Reflective Journaling Intervention
Brief Title: Does a Novel Intervention Targeting Derailment Decrease Depressive Symptoms?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB0148200
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Depression; Depressive Symptoms; Derailment; Anxiety
Keywords: Depression; Identity Continuity; Randomized Control Trial; Journaling
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Investigators will utilize a single-blind approach where participants will not be made aware of the purpose of the intervention. Participants in both arms will be told that the purpose of the study is "to determine the efficacy of a novel five-session journaling intervention, which explores concepts related to self-continuity". This is partly true for those in the experimental arm. The main purpose of the study is twofold: (1) to explore the efficacy of the experimental journaling intervention's in reducing levels of derailment and (2) to test the hypothesis that decreasing derailment- a temporal discordance of the self- will lead to a decrease in depressive symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Derailment-Focused Reflective Journaling Condition (Experimental): Participants will be tasked with engaging in a 5-session journaling intervention where participants reflect on core aspects about their (participants') selves within traditional developmental stages (e.g., first semester in college, early childhood, etc.).
  Interventions: Behavioral: Derailment-Focused Reflective Journaling
- Everyday Tasks Reflective Journaling Condition (Placebo Comparator): Participants will be tasked with engaging in a 5-session journaling intervention where they (participants) reflect on everyday tasks (e.g., their last trip to the grocery store, the last movie they saw, etc.).
  Interventions: Other: Everyday Tasks Reflective Journaling

INTERVENTIONS:
Behavioral: Derailment-Focused Reflective Journaling — Experimental group aimed at decreasing anxiety symptoms
  Arms: Derailment-Focused Reflective Journaling Condition
Other: Everyday Tasks Reflective Journaling — Control group
  Arms: Everyday Tasks Reflective Journaling Condition

SUMMARY:
The goal of this clinical trial is to explore the efficacy of a reflective journaling intervention-"Me Through Time"- in decreasing levels of derailment, and its impact on downstream depressive symptoms.

DETAILED DESCRIPTION:
The population will consist of those who: are considered as emergent adults (18-29 years) with at least moderate to severe depressive symptoms (a score of at least 20 on the BDI-II), moderate anxiety symptoms (a score of at least 10 on the GAD-7), and high levels of derailment (a score of at least 37 on the Derailment Scale).

Main research questions are as follows:

* Does the "Me Through Time" journaling intervention predict decreased derailment and depressive symptoms at post-assessment compared to the severity of pre-assessment derailment and depressive symptoms?
* Are post-assessment derailment and depressive symptoms lower for those who engaged in the "Me Through Time" journaling intervention compared to a control journaling intervention?

Participants will be asked to complete structured journal entries over the course of 5 sessions over 2 weeks, whereby each session addresses a different critical time period. These include: (1) first semester of college, (2) high school years, (3) middle school years, (4) early childhood, and finally (5) desired future. Participants will also be tasked with completing several assessment scales both before and after completing the "Me Through Time" journaling experience, as well as at the midway point.

The investigators will compare an experimental group engaging in the novel, derailment-focused "Me Through Time" journaling intervention with a control group engaging in a neutral, non-identity-based reflective journaling activity spanning the same time period as the "Me Through Time" intervention to see if post-assessment derailment and depressive symptoms are lower for those who engaged in the "Me Through Time" journaling intervention compared to the control journaling intervention.

The investigators hypothesize that those in the experimental condition will endorse significantly lower derailment and depressive symptoms at T2 than those in the control condition. Further, the investigators hypothesize significant decreases in T1 to T2 depressive symptoms and derailment for those in the experimental condition, but not in the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged 18-29.
* Participants must be fluent in English.
* Participants must have attended at least one semester of college.
* Participants must live in the United States
* Participants must have a score on the Derailment Scale of at least 37 at pre-assessment.
* Participants must have a score on the Beck Depression Inventory II of at least 20 at pre- assessment.
* Participants must have a score on the GAD-7 of at least 10 at pre-assessment.
* Participants must be willing and able to engage in a 2-week reflective journaling experience.

Exclusion Criteria:

* Those outside of the specified age range.
* Those who are not fluent in English.
* Those who have not attended at least one semester of college.
* Those who do not live in the United States.
* Those who have a score on the Derailment Scale of less than 37 at pre-assessment.
* Those have a score on the Beck Depression Inventory II of less than 20 at pre- assessment.
* Those who have a score on the GAD-7 of less than 10 at pre-assessment.
* Those who are neither willing nor able to engage in a 2-week reflective journaling experience.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Change from Pre-Assessment in Depressive Symptoms on the Beck Depression Inventory II (BDI-II) at Week 2 (Session 6/Post-Assessment) | Baseline (Pre-Assessment) and Week 2 (Session 6/Post-Assessment)
  The Beck Depression Inventory II is a validated, 21-item self-reported instrument assessing the severity of depression symptomatology in adolescents and adults. Items are summed to create a total score, whereby higher scores indicate higher levels of depressive symptoms. Scores range from 0-63, and a total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Change from Pre-Assessment in Levels of Derailment on the Derailment Scale at Session 5 | Pre-Assessment (Baseline) and Session 5
  The Derailment Scale is a validated, 10-item self-reported instrument that measures one's level of derailment - that is, one's perceptions of global change in self and direction. Possible scores range from 10-50, whereby higher scores indicate higher levels of derailment.

SECONDARY OUTCOMES:
Change from Pre-Assessment in Anxiety Symptoms on the Generalized Anxiety Disorder - 7 (GAD-7) at Week 2 (Session 6/Post-Assessment) | Baseline (Pre-Assessment) and Week 2 (Session 6/Post-Assessment)
  The Generalized Anxiety Disorder 7-item is a validated, self-reported instrument that is used to assess symptoms of anxiety based on the generalized anxiety disorder diagnostic criteria described in the Diagnostic and Statistical Manual of Mental Disorders. Possible scores range from 0 to 21, whereby higher score indicate higher levels of anxiety symptoms. Specifically, a raw score of 0-4 is considered minimal range, 5-9 is mild, 10-14 is moderate, and 15-21 is severe.
Change from Pre-Assessment in Levels of Positive and Negative Affect on the Positive and Negative Affect Schedule (PANAS) at Week 2 (Session 6/Post-Assessment) | Baseline (Pre-Assessment) and Week 2 (Session 6/Post-Assessment)
  The Positive and Negative Affect Schedule is a validated, self-reported instrument that is used to measure mood and emotion, specifically positive affect and negative affect. It contains 20 items, 10 of which measure positive affect (e.g., excited, inspired) and the other 10 of which measure negative affect (e.g., upset, afraid). One's score on this instrument is separated into Positive Affect and Negative Affect scores, with a higher score indicating more positive or negative affect, respectively. Scores for both Positive Affect and Negative Affect Scores can range from 10-50.
Change from Pre-Assessment in Levels of Perceived Stress on the Perceived Stress Scale (PSS) at Week 2 (Session 6/Post-Assessment) | Baseline (Pre-Assessment) and Week 2 (Session 6/Post-Assessment)
  The Perceived Stress Scale is a validated, 10-item self-reported instrument that measures the perception of stress; that is, it is a measure of the degree to which situations in one's life are appraised as stressful. Possible scores range from 0-40, with higher scores representing higher levels of stress.
Change from Pre-Assessment in Levels of Optimism Versus Pessimism on the Life Orientation Test - Revised (LOT - Revised) at Week 2 (Session 6/Post-Assessment | Baseline (Pre-Assessment) and Week 2 (Session 6/Post-Assessment)
  The Life Orientation Test - Revised is a validated, 10-item self-reported instrument that is used to measure individual differences in optimism versus pessimism. Negatively worded items (Items 3, 7, and 9) are reverse coded before scoring. Responses to these items are then summed with the participant's responses to Items 1, 4, and 10 to compute an overall optimism score. Items 2, 5, 6, and 8 are fillers and should not be scored. Thus, scores on this instrument range from 0 to 24, whereby lower scores indicate lower optimism (higher pessimism) and higher scores indicate higher optimism (lower pessimism).

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No